CLINICAL TRIAL: NCT06387550
Title: Effects of Eccentric Training on Glycemic Control and Quality of Life in Patients With Type II Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/3
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Type II Diabetes Mellitus
Keywords: Eccentric training, Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a pre-post quasi experimental study having one group analysis.Participants will be selected through inclusion and exclusion criteria then pre assessment would be done that include HBA1C and EQ5DL QOL tool, followed by intervention and post assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eccentric Training Group (Experimental): Patients in this group firstly passing through warm up phase that include hip circles and shoulder rolls(1 sets of 5 reps), participants are trained on bicycle ergometer for 15 minutes on 2-3 times a week and its duration is increased according to patient tolerance, after that they will be pass through exercise phase that include squating, lunges and leg press (8-10 reps of 3 sets) after that cool down phase begin that include cat cow stretch and oblique stretch (5 reps of 1 set)
  Interventions: Procedure: Eccentric Training

INTERVENTIONS:
Procedure: Eccentric Training — Warm up phase that include hip circles and shoulder rolls(1 sets of 5 reps), participants are trained on bicycle ergometer for 15 minutes on 2-3 times a week and its duration is increased according to patient tolerance, after that they will be pass through exercise phase that include squating, lunges and leg press (8-10 reps of 3 sets) after that cool down phase begin that include cat cow stretch and oblique stretch (5 reps of 1 set)

SUMMARY:
Diabetes is defined by the level of hyperglycemia its a metabolic chronic disorder that furthur lead to life threatning medical conditions however, the prevalence of diabetes is rapidly increasing day by day in both developed and developing countries making it global pandemic and type II is more prevalent. Life dependency is increased due to long term effects of diabetes in specifically older individuals. Physical activity and exercise improves glucose tolerance and also reduces other life threatening diabetic complications, improving the quality of life in diabetic population.

DETAILED DESCRIPTION:
Diabetes is a metabolic chronic disorder and its becoming a global pandemic and its prevalence rises quickly in both developed and developing countries.Diabetes confirmation is done through levels of hyperglycemia. According to American Diabetic Association level of HBA1C is greater than 6.4

% indicate presence of diabetes.Type II is more prevalent and its deteriorting effect on body with increasing age are more pronounced.Insuline resistance and impaired glucose tolerance are seen in type II diabetes mellitus patients.

Studies depict that regular exercise improve glycemic control and improve insuline sensitivity and enhance glucose uptake by muscles.

Strength training enhance quality of life and protect your joints from injury. Previous studies have specified the impact of several types of training on older adults, young healthy adults and diabetic patients but there is limited literature found in terms of solely observing the effect of eccentric training on glycemic control and quality of life in diabetic patient.

Current study was designed to determine the effects of eccentric training on glycemic control and quality of life in type II diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Blood pressure should be <140/90mm of Hg
* Diagnosed Diabetic patient (HBA1C>6.4%)
* Adults (Age 40 +) from Rawalpindi and Islamabad

Exclusion Criteria:

* Acute infection
* History of recent trauma
* Acute coronary syndrome
* Peripheral vascular diseases

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | 8 weeks
  Lab investigation of glycemic control will be through HBA1C test.
Patient's quality of life | 8 weeks
  Quality of life will be assessed using EQ5DL Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan